CLINICAL TRIAL: NCT04321486
Title: Natural History and Patient Journey in Dementia: a Nationwide Linked Electronic Health Records Study of 5.6 Million Individuals.
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Other Study IDs: ISAC18_228
Record Dates: First submitted 2020-03-23; First posted 2020-03-25 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-03

CONDITIONS: Dementia, Alzheimer, Electronic Health Records, Hospitalizations, Epidemiology, Comorbidity, United Kingdom, Incidence, Mortality, Cause of Death
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: The study does not have an intervention, but observe the dementia incidence of the UK disease-free population. — The study does not have an intervention, but observe the dementia incidence of the UK disease-free population.

SUMMARY:
The trajectory of dementia patients within the national health system and their recent temporal trends remains to be fully elucidated. To study the dementia incidence, mortality and case-fatality, we implemented a longitudinal cohort study with the linked electronic health records of 5.6 million population in the UK from 1998 to 2016 (CALIBER). A matched case-control study design was used to investigate the causes of hospitalization and death comparing individuals with and without incident dementia.

ELIGIBILITY:
Inclusion Criteria:

* We identify individuals aged 30 years or older and registered in the current primary care practice for at least one year.

Exclusion Criteria:

* Individuals are excluded if they had a prior history of dementia before study entry.

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We implement two study designs, first a longitudinal cohort study to assess dementia incidence and second a matched case-control study for mortality, cause of death and hospitalization.
  We identify individuals aged 30 years or older and registered in the current primary care practice for at least one year. Individuals are excluded if they had a prior history of dementia before study entry. For the nested case-control study, controls are matched to incident dementia patients according to sex and age (10-year age strata).
Sampling Method: Non-Probability Sample
Enrollment: 4309481 (Actual)
Dates: Start 1998-01-01 (Actual); Primary Completion 2016-05-31 (Actual); Study Completion 2020-11-30 (Estimated)

PRIMARY OUTCOMES:
Incidence and mortality of dementia | Jan 1st 1998 - May 31st 2016